CLINICAL TRIAL: NCT01253954
Title: Epidemiology of Invasive Candida Infections in Critically Ill Patients: A Multicenter, Prospective, Observational Study in China
Brief Title: A Multicenter Observational Study of Invasive Candida Infections Among ICU Patients in China
Acronym: china-scan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Collaborators: QLT Inc. (Industry)
Responsible Party: Haibo Qiu, Southeast University
Other Study IDs: 1234
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2009-11

CONDITIONS: Candidiasis
Keywords: invasive candida infection
MeSH Terms: conditions — Candidiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU patients with IFI: 1

SUMMARY:
The incidence of invasive candida infection (ICI) in critically ill patients is increasing day by day. The crude mortality of IFI in ICU could be as high as 25%-75% depending on their age, underlying conditions, and so on. Candida albicans was by far the predominant species in most countries, causing up to two thirds of all cases of invasive candidiasis. However, a shift toward non-albicans Candida species has been observed. Although the studies of ICI cause universal attention recently, there is still no large-scale, multi-center epidemiological research in China focusing on ICI in critically ill patients, therefore we conducted a large-scale multi-center observational study of IFI in critically ill patients named "China Scan" (CHINA Survey of Candidiasis in ICU) to assess the current incidence, mortality, pathogen spectrum, management, and risk factors for ICI in China ICUs.

DETAILED DESCRIPTION:
Background of the study:

The incidence of invasive candida infection (ICI) in critically ill patients is increasing day by day. The crude mortality of ICI in ICU could be as high as 25%-75% depending on their age, underlying conditions, and so on. Candida albicans was by far the predominant species in most countries, causing up to two thirds of all cases of invasive candidiasis. However, a shift toward non-albicans Candida species has been observed. Although the studies of ICI cause universal attention recently, there is still no large-scale, multi-center epidemiological research in China focusing on IFI in critically ill patients, therefore we conducted a large-scale multi-center observational study of IFI in critically ill patients named "China Scan" (CHINA Survey of Candidiasis in ICU) to assess the current incidence, mortality, pathogen spectrum, management, and risk factors for ICI in China ICUs.

Objective of the study:

Determine the current incidence of IFI in ICUs in China. Describe the risk factors for IFI in China ICUs. Explore the pathogen spectrum of IFI in ICUs in China. Describe the in vitro antifungal susceptibility of Candida isolates. Describe the antifungal treatment for ICU patients with IFI. Evaluate in-hospital mortality among patients with IFI in ICUs.

ELIGIBILITY:
Inclusion criteria:

-Adult ICU patients above 18 with ICI-

Exclusion criteria:

-Non ICI-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU patients above 18 with invasive candida infection
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Determine the current incidence and in-hospital mortality of invasive candidas infection in ICUs in China. | 300 charactors

SECONDARY OUTCOMES:
Describe the risk factors for ICI in China ICUs. Explore the pathogen spectrum of ICI in ICUs in China. Describe the in vitro antifungal susceptibility of Candida isolates. Describe the antifungal treatment for ICU patients with ICI. | 300 charactors

CONTACTS AND LOCATIONS:
Locations (1):
- Gulou District, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Cui N, Wang H, Su L, Qiu H, Li R, Liu D; China-SCAN Team. Initial therapeutic strategy of invasive candidiasis for intensive care unit patients: a retrospective analysis from the China-SCAN study. BMC Infect Dis. 2017 Jan 23;17(1):93. doi: 10.1186/s12879-017-2207-1. PMID 28114898
- [Derived] Guo F, Yang Y, Kang Y, Zang B, Cui W, Qin B, Qin Y, Fang Q, Qin T, Jiang D, Li W, Gu Q, Zhao H, Liu D, Guan X, Li J, Ma X, Yu K, Chan D, Yan J, Tang Y, Liu W, Li R, Qiu H; China-SCAN Team. Invasive candidiasis in intensive care units in China: a multicentre prospective observational study. J Antimicrob Chemother. 2013 Jul;68(7):1660-8. doi: 10.1093/jac/dkt083. Epub 2013 Mar 29. PMID 23543609